CLINICAL TRIAL: NCT03636373
Title: Investigator-Initiated, Pilot Study Evaluating The Efficacy Of Etanercept In Acute Gout
Brief Title: Pilot Study Evaluating The Efficacy Of Etanercept In Acute Gout
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The Sponsor has decided to stop funding this study due to lack of enrollment during COVID-19 pandemic and decreased interest in funding investigator initiated studies pertaining to the study drug
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Naomi Schlesinger, MD, Professor of Medicine, Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro2018000562
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Gout Attack
MeSH Terms: interventions — Etanercept; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Subjects will be administered a single dose of etanercept 50 mg subcutaneously (SC), at the onset of an acute gout attack, or a single dose of triamcinolone acetonide 40 mg intramuscularly (IM)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etanercept (Experimental): Subjects will be administered etanercept 50 mg subcutaneously and a placebo intramuscularly
  Interventions: Drug: Etanercept
- Triamcinolone acetonide (Active Comparator): Subjects will be administered triamcinolone acetonide 40 mg intramuscularly and a placebo subcutaneously
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Etanercept — Subjects will receive 50 mg of study drug on visit 1. A second dose of study drug will be administered if the pain intensity is ≥ 5 on a pain scale of 0-10 at Visit 2
  Arms: Etanercept
Drug: Triamcinolone Acetonide — Subjects will be administered triamcinolone acetonide 40 mg intramuscularly on visit 1. A second dose of drug will be administered if the pain intensity is ≥ 5 on a pain scale of 0-10 at Visit 2
  Arms: Triamcinolone acetonide

SUMMARY:
The purpose of this pilot study is to investigate the safety and efficacy of etanercept (Enbrel™; Amgen) for the treatment of an acute gout attack will be non-inferior to triamcinolone acetonide an FDA approved drug to treat acute gout attacks.

DETAILED DESCRIPTION:
The study was designed as a 14-day, two center- pilot randomized, active-controlled, double-blind, study. The study was approved by the Institutional Review Board (IRB) Pro2018000562. Patients were screened for eligibility at the time of an acute flare. Patients aged 28-55 years with an acute gout flare meeting the validated definition of flare were enrolled (12). Onset of current acute gout flare was within 3 days prior to randomization and baseline pain intensity ≥50 mm on a 0-100 mm visual analogue scale (VAS), Gout patients were defined by a confirmed diagnosis of crystal proven gout and or a score of ≥ 8 on the 2015 American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) Gout Classification Criteria (13).

Patients recorded pain intensity in the most affected joint prior to treatment. Efficacy, including pain on a 0-100 mm VAS, and safety assessments were conducted at 24 and 72 hours, 7 and 14 days after baseline.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients age ≥18 to ≤85 year
2. History of established gout
3. Onset of current acute gout attack within 4 days prior to randomization with: presence of any warm joint, swollen joint, pain score at rest ≥5 on the 0-10 pain scale, patient self-report of acute gout attack
4. Baseline pain intensity ≥5 on a 0-10 pain scale;
5. Tender (≥1 on a 0-4-point Likert scale) and swollen (≥1 on a 0-4-point Likert scale) index joint;
6. If on urate-lowering therapy, a stable dose and regimen for at least 2 weeks prior to randomization, and expectance to remain on a stable dose and regimen for the duration of the double-blind treatment period, and;
7. Body mass index (BMI) ≤45 kg/m2.

Exclusion Criteria:

1. Use of intra-articular or IM corticosteroids within 14 days prior to screening;
2. Use of an IL-1 inhibitor, TNF inhibitor or other biologic or investigational drug within 30 days prior to screening;
3. History of a drug allergy to either study drug;
4. Diagnosis or history of:

   1. rheumatoid arthritis (RA);
   2. infectious/septic or other inflammatory arthritis;
   3. alcoholic hepatitis or nonalcoholic steatohepatitis;
   4. immunodeficiency syndromes, including Human Immunodeficiency Virus (HIV) infection;
   5. Stage IIIb, IV, or V chronic kidney disease;
   6. idiopathic thrombocytopenic purpura;
   7. active, severe chronic pulmonary disease (eg, requiring oxygen therapy);
   8. uncontrolled hypertension (≥ 200/105 mmHg);
   9. symptomatic (New York Heart Association Class II, III, or IV) congestive heart failure;
   10. uncontrolled diabetes Type I or II (recent blood glucose > 300 mg/dL);
   11. myocardial infarction, unstable cardiac arrhythmias or unstable symptomatic coronary ischemia, within the past 12 months before randomization;
   12. history of malignancy of any organ system within the past 5 years;
   13. multiple sclerosis or any other demyelinating disease, or;
   14. major chronic inflammatory disease or connective tissue disease other than RA or psoriatic arthritis (PsA), including but not limited to fibromyalgia or systemic lupus erythematosus (with the exception of secondary Sjögrens syndrome, etc.);
5. Contraindication to IM injection;
6. Donation or loss of ≥400 milliliters (mL) of blood in the 8 weeks before dosing;
7. Any live vaccination in the 3 months before the start of the study;
8. Active infection (including chronic or localized infections) for which antiinfectives were indicated within 4 weeks before screening;
9. Any serious infection, defined as requiring hospitalization or intravenous anti-infectives, within 8 weeks before first dose of investigational product;
10. Prosthetic joint infection within 5 years of screening, or native joint infection within 1 year of screening;
11. Known alcohol addiction or dependency, daily alcohol use, or current substance use or abuse;
12. Positive medical history for hepatitis B or C (subjects with a history of hepatitis B vaccination without history of hepatitis B infection are allowed to enroll);
13. History of active tuberculosis;
14. Positive test for tuberculosis during screening, defined as positive Purified Protein Derivative (PPD) skin test (≥5 mm induration at 48-72 hours after test is placed), or positive Quantiferon test;
15. Pregnant or nursing (lactating) women
16. Female patients who are physiologically capable of becoming pregnant must use an acceptable method of contraception

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Schlesinger, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School/ Rutgers RWJMS Gout center
Locations (1):
- Rutgers, Robert Wood Johnson Medical School, Clinical Research Center, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Subjects will be administered etanercept 50 mg subcutaneously and a placebo intramuscularly
  Etanercept: Subjects will receive 50 mg of study drug on visit 1. A second dose of study drug will be administered if the pain intensity is ≥ 5 on a Visual Analog Scale (VAS) of 0-10 at Visit 2
- Triamcinolone Acetonide: Subjects will be administered triamcinolone acetonide 40 mg intramuscularly and a placebo subcutaneously
  Triamcinolone Acetonide: Subjects will be administered triamcinolone acetonide 40 mg intramuscularly on visit 1. A second dose of drug will be administered if the pain intensity is ≥ 5 on a Visual Analog Scale (VAS) of 0-10 at Visit 2
Period: Overall Study
Arm/Group | Etanercept | Triamcinolone Acetonide
Started | 3 | 2
Completed | 2 | 2
Not Completed | 1 | 0
Not completed — Study closure due to Covid-19 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Etanercept: Subjects will be administered etanercept 50 mg subcutaneously and a placebo intramuscularly
  Etanercept: Subjects will receive 50 mg of study drug on visit 1. A second dose of study drug will be administered if the pain intensity is ≥ 5 on a Visual Analog Scale (VAS) of 0-10 at Visit 2 with 0 indicating no pain and 10 indicating intense pain.
- Triamcinolone Acetonide: Subjects will be administered triamcinolone acetonide 40 mg intramuscularly and a placebo subcutaneously
  Triamcinolone Acetonide: Subjects will be administered triamcinolone acetonide 40 mg intramuscularly on visit 1. A second dose of drug will be administered if the pain intensity is ≥ 5 on a Visual Analog Scale (VAS) of 0-10 at Visit 2 with 0 indicating no pain and 10 indicating intense pain.
- Total: Total of all reporting groups
Arm/Group | Etanercept | Triamcinolone Acetonide | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Patient reported pain [Mean (Full Range); unit: units on a scale] — Visual Analog Scale used to measure severity of gout pain in the target joint at screening, visit 2, visit 3 and visit 4. Patient reported pain score 0 indicates no pain (better outcome) and 10 indicates severe pain (worse outcome).
  Baseline patient reported pain mean score Etanercept Arm {( 8 + 8 + 7) / 3} = 7.67 Triamcinolone Acetonide Arm {( 5+7) /2} = 6; Total for both arms {(8+8+7+5+7= 35)/5) =7
  units on a scale | 7.67 [7 to 8] | 6.00 [5 to 7] | 7.00 [5 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Joint Pain Intensity in the Most Affected Joint
Description: Pain intensity in the most affected baseline joint measured by the numeric 0-10 Visual Analog Scale at 72 hours with 0 indicating no pain and 10 indicating intense pain. Higher score indicating a worse outcome.
Time Frame: 72 hours
Population: Evaluate the efficacy of etanercept, compared to triamcinolone acetonide in patients with acute gout attack
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Etanercept: Subjects will be administered etanercept 50 mg subcutaneously and a placebo intramuscularly
  Etanercept: Subjects will receive 50 mg of study drug on visit 1. A second dose of study drug will be administered if the pain intensity is ≥ 5 on a Visual Analog Scale of 0-10 at Visit 2 with 0 indicating no pain and 10 indicating intense pain. Higher score indicating a worse outcome.
- Triamcinolone Acetonide: Subjects will be administered triamcinolone acetonide 40 mg intramuscularly and a placebo subcutaneously
  Triamcinolone Acetonide: Subjects will be administered triamcinolone acetonide 40 mg intramuscularly on visit 1. A second dose of drug will be administered if the pain intensity is ≥ 5 on a Visual Analog Scale of 0-10 at Visit 2 with 0 indicating no pain and 10 indicating intense pain. Higher score indicating a worse outcome.
Arm/Group | Etanercept | Triamcinolone Acetonide
Number analyzed (Participants) | 3 | 2
score on a scale | 5 [0 to 8] | 1.5 [0 to 3]
Statistical Analysis 1: Comparison: Etanercept vs Triamcinolone Acetonide; Mean Outcome measure Etanercept arm { ( 8 + 0 + 7)/3 = 5} Triamcinolone Arm { (3+0) /2 = 1.5 }; Test type: Non-Inferiority — On a 10 point Likert Pain Scale, non-inferiority margin for the difference is 1.04. Using a Student t-test, there was 80% power for the difference in pain levels to exceed -1.04; p = 1.00, t-test, 1 sided

2. Secondary Outcome: Joint Pain on Numeric Pain Scale
Description: Patient's assessment of joint pain intensity in the most affected baseline joint on a numeric 0-10 Visual Analog Scale at Baseline and post-dose Days with 0 indicating no pain and 10 indicating intense pain. Higher score indicating a worse outcome.
Time Frame: Baseline, Days 4, 7, and 14
Population: 2 patients were enrolled in Triamcinolone acetonide arm and 3 patients were enrolled in Etanercept arm. However only two patients in the Etanercept arm completed the study. One patient completed only 2 study visits since the study was put on hold due to COVID-19 pandemic.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Triamcinolone Acetonide: Subjects will be administered Triamcinolone acetonide 40 mg intramuscularly and a placebo subcutaneously
  Triamcinolone Acetonide: Subjects will be administered triamcinolone acetonide 40 mg intramuscularly on visit 1. A second dose of drug will be administered if the pain intensity is ≥ 5 on a pain scale of 0-10 at Visit 2
  Two patients were randomly assigned to the TA arm.
- Etanercept: Subjects will be administered Etanercept 50 mg subcutaneously and a placebo intramuscularly
  Etanercept: Subjects will receive 50 mg of study drug on visit 1. A second dose of study drug will be administered if the pain intensity is ≥ 5 on a pain scale of 0-10 at Visit 2
  Three patients were randomly assigned to the etanercept arm.
Arm/Group | Triamcinolone Acetonide | Etanercept
Number analyzed (Participants) | 2 | 3
score on a scale
  Visit 1 (Baseline) | 6 [5 to 7] | 7.67 [7 to 8]
  Visit 2 (Day 4) | 1.5 [0 to 3] | 5 [0 to 8]
  Visit 3 (Day 7): number analyzed (Participants) | 2 | 2
  Visit 3 (Day 7) | 1 [0 to 2] | 3 [0 to 6]
  Visit 4 (Day 14): number analyzed (Participants) | 2 | 2
  Visit 4 (Day 14) | 1 [0 to 2] | 0.5 [0 to 1]
Statistical Analysis 1: Comparison: Triamcinolone Acetonide vs Etanercept; Test type: Superiority; p = 1.00, t-test, 2 sided

3. Secondary Outcome: Patient's Assessment of Response to Treatment
Description: Patient's global assessment of response to treatment (Likert), options are None, Poor, Acceptable, Good, Excellent
Time Frame: Day 4, 7 and 14
Population: 4 subjects completed the study with 2 in each arm. Additionally, 1 more subject completed 2 visits (Day 1 and Day 4) only 2 visits in Etanercept arm. Therefore, 2 subjects in Triamcinolone acetonide completed Visit 2 while 3 subjects in Etanercept arm completed this Visit. However, out of the 2 participants who completed all study visits in the Etanercept arm, only 1 participant completed "Patient's assessment of response to treatment." Thus, only 1 participant was included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone Acetonide | Etanercept
Number analyzed (Participants) | 2 | 3
Participants
  Visit 2 (Day 4): None | 0 | 1
  Visit 2 (Day 4): Poor | 0 | 0
  Visit 2 (Day 4): Acceptable | 0 | 0
  Visit 2 (Day 4): Good | 2 | 1
  Visit 2 (Day 4): Excellent | 0 | 1
  Visit 3 (Day 7): number analyzed (Participants) | 2 | 2
  Visit 3 (Day 7): None | 0 | 0
  Visit 3 (Day 7): Poor | 0 | 1
  Visit 3 (Day 7): Acceptable | 0 | 0
  Visit 3 (Day 7): Good | 0 | 0
  Visit 3 (Day 7): Excellent | 2 | 1
  Visit 4 (Day 14): number analyzed (Participants) | 2 | 1
  Visit 4 (Day 14): None | 0 | 0
  Visit 4 (Day 14): Poor | 0 | 1
  Visit 4 (Day 14): Acceptable | 0 | 0
  Visit 4 (Day 14): Good | 1 | 0
  Visit 4 (Day 14): Excellent | 1 | 0
Statistical Analysis 1: Comparison: Triamcinolone Acetonide vs Etanercept; Test type: Superiority; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Physician's Assessment of Response to Treatment
Description: Physician's global assessment of response to treatment None, Poor, Acceptable, Good, Excellent
Time Frame: Post-dose days 4, 7 and 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone Acetonide | Etanercept
Number analyzed (Participants) | 2 | 3
Participants
  Visit 2 (Day 4): None | 0 | 1
  Visit 2 (Day 4): Poor | 0 | 0
  Visit 2 (Day 4): Acceptable | 0 | 0
  Visit 2 (Day 4): Good | 1 | 2
  Visit 2 (Day 4): Excellent | 1 | 0
  Visit 3 (Day 7): number analyzed (Participants) | 2 | 2
  Visit 3 (Day 7): None | 0 | 0
  Visit 3 (Day 7): Poor | 0 | 0
  Visit 3 (Day 7): Acceptable | 0 | 1
  Visit 3 (Day 7): Good | 0 | 0
  Visit 3 (Day 7): Excellent | 2 | 1
  Visit 4 (Day 14): number analyzed (Participants) | 2 | 2
  Visit 4 (Day 14): None | 0 | 0
  Visit 4 (Day 14): Poor | 0 | 0
  Visit 4 (Day 14): Acceptable | 0 | 0
  Visit 4 (Day 14): Good | 0 | 1
  Visit 4 (Day 14): Excellent | 2 | 1
Statistical Analysis 1: Comparison: Triamcinolone Acetonide vs Etanercept; Test type: Superiority; p = 0.05, t-test, 2 sided

5. Secondary Outcome: Rescue Medication
Description: Total number of patients taking rescue medication after the administration of study medication while on study.
  Compare the use of rescue medication in etanercept and triamcinolone acetonide patients: for those patients having difficulty tolerating their pain, despite the treatment, were allowed to take rescue medication for pain. A paper diary was given to each patient at baseline visit to record the rescue medications.
Time Frame: Day 1 (Baseline visit - Visit 1) through Day 14 (Visit 4).
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone Acetonide | Etanercept
Number analyzed (Participants) | 2 | 3
Participants
  Used Rescue Medications | 1 | 2
  Did not use Rescue Medications | 1 | 1
Statistical Analysis 1: Comparison: Triamcinolone Acetonide vs Etanercept; Test type: Superiority; p = 0.05, t-test, 2 sided

6. Secondary Outcome: Safety and Tolerability of Etanercept
Description: Safety and tolerability as assessed by subjects with adverse events and serious adverse events from baseline through Visit 5 safety follow-up
Time Frame: Day 1 (Baseline visit - Visit 1) through Day 30 (Safety follow up phone visit -Visit 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone Acetonide | Etanercept
Number analyzed (Participants) | 2 | 3
Participants
  Reported Adverse Events | 1 | 1
  Did not report Adverse Events | 1 | 2
Statistical Analysis 1: Comparison: Triamcinolone Acetonide vs Etanercept; Test type: Superiority; p = 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse event related information was collected at baseline, visit 2, 3 and 4 and the phone call at the end of the study period (~30 days)
Arm/Group | Etanercept | Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=3) | Triamcinolone Acetonide (N=2)
Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Swelling right peri-achilles area
Fatigue (General disorders) | 0 (0) | 1 (1)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03636373/Prot_003.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03636373/SAP_004.pdf
  • Informed Consent Form (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03636373/ICF_005.pdf